CLINICAL TRIAL: NCT06808490
Title: Exercise and Endocannabinoids for Brain and Mental Health
Acronym: EMBH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wayne State University (Other)
Responsible Party: Principal Investigator, Hilary Marusak, Associate Professor, Wayne State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: IRB-21-04-3502
Record Dates: First submitted 2025-01-07; First posted 2025-02-05 (Actual); Last update posted 2025-02-05 (Actual); Status verified 2025-01

CONDITIONS: Children; Adolescents
Keywords: Exercise; Endocannabinoid; Anxiety; Meditation; Stretching
MeSH Terms: conditions — Motor Activity; Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Moderate Intensity Exercise (Experimental)
  Interventions: Behavioral: Moderate Intensity Exercise
- Light Intensity Stretching (Active Comparator)
  Interventions: Behavioral: Light Intensity Stretching
- Seated Meditation (Active Comparator)
  Interventions: Behavioral: Seated Meditation

INTERVENTIONS:
Behavioral: Moderate Intensity Exercise — Participants randomized to the moderate intensity exercise condition will complete a 30 min session on a motor driven treadmill. Participants will complete a 3-minute warm-up at low speed on a treadmill. Speed and incline will be increased in 3-minute increments until moderate-intensity exercise, defined as the goal of participants staying within a target zone of 50-70% AAMHR while briskly walking and/or jogging depending on current fitness status.
  Arms: Moderate Intensity Exercise
Behavioral: Light Intensity Stretching — Participants randomized into the light stretching condition will complete a 30-minute video, tailored for 9-17-year-olds. This video leads participants through a series of seated arm, torso, leg, knee and shoulder stretches on a yoga mat. Participants will be monitored throughout the stretching session by a trained research assistant, and HR and perceived exertion will also be measured throughout. The research assistant may make modifications to the poses in real-time to ensure that AAMHR is kept below 40%.
  Arms: Light Intensity Stretching
Behavioral: Seated Meditation — Participants randomized into the meditation condition will complete a 30-minute video, tailored for 9-17-year-olds. This video leads participants through a seated guided meditation on a yoga mat. This includes a series of breathing, visualization, and body awareness exercises. Participants will be monitored throughout the meditation session by a trained research assistant, and HR and perceived exertion will also be measured throughout, to ensure that AAMHR is kept below 30%.
  Arms: Seated Meditation

SUMMARY:
This study will explore how exercise affects brain chemicals called endocannabinoids, which may improve thinking skills and reduce feelings of stress, anxiety, and low mood in children and teens aged 9 to 17. Participants will take part in a single 30-minute activity session, where they will be randomly assigned to one of three groups:

1. Moderate-intensity exercise (walking or running on a treadmill at 50-70% of their maximum heart rate).
2. Light stretching (gentle movements at less than 40% of their maximum heart rate).
3. Seated meditation (relaxing without movement at less than 30% of their maximum heart rate).

The investigators will measure endocannabinoid levels, thinking skills, and mood before and after the activity to see how these activities affect the brain and emotions.

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed and dated informed consent form
* Stated willingness to comply with all study procedures and available for the duration of the study
* 9-17 years of age
* Adolescent and parent/guardian are English-speaking, as study assessments are in English
* Right-handed

Exclusion Criteria:

* Head injury
* Sensory (e.g., hearing) impairment
* Physical (e.g., motor, balance) impairment
* Physical disabilities
* Neurological disorders
* Any condition that would contraindicate blood draws

Ages: 9 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 68 (Actual)
Dates: Start 2021-12-21 (Actual); Primary Completion 2024-03-18 (Actual); Study Completion 2024-03-18 (Actual)

PRIMARY OUTCOMES:
Endocannabinoid (eCB) Concentrations | Within 30 minutes before and after exercise or control conditions
  Plasma and saliva samples will be collected immediately before and after exercise or control conditions. Samples will be analyzed using liquid chromatography-mass spectrometry to quantify concentrations of eCBs.
Cognitive performance (Dimensional Change Card Sort Test) | Within 30 minutes before and after exercise or control conditions
  The NIH Toolbox® iPad application will be administered to measure executive functioning before and after the exercise or control condition: Dimensional Change Card Sort Test (DCCS).
Cognitive performance (Flanker Inhibitory Control and Attention Test) | Within 30 minutes before and after exercise or control conditions
  The NIH Toolbox® iPad application will be administered to measure executive functioning before and after the exercise or control condition: Flanker Inhibitory Control and Attention Test (Flanker).
Cognitive performance (Pattern Comparison Processing Speed Test) | Within 30 minutes before and after exercise or control conditions
  The NIH Toolbox® iPad application will be administered to measure executive functioning before and after the exercise or control condition: Pattern Comparison Processing Speed Test (PCT).
Cognitive performance (Picture Sequence Memory Test) | Within 30 minutes before and after exercise or control conditions
  The NIH Toolbox® iPad application will be administered to measure executive functioning before and after the exercise or control condition: Picture Sequence Memory Test (PSMT).
Anxiety symptoms | Within 30 minutes before and after exercise or control conditions
  State-Trait Anxiety Inventory for children
Affect | Within 30 minutes before and after exercise or control conditions
  Positive and Negative Affect Schedule (PANAS) - Child Version
Mood state | Within 30 minutes before and after exercise or control conditions
  Mood and Feelings Questionnaire for Children

CONTACTS AND LOCATIONS:
Overall Officials: Hilary Marusak, Principal Investigator — Wayne State University; Jeanne Barcelona, Principal Investigator — Wayne State University
Locations (1):
- Tolan Park Medical Building, Detroit, Michigan, United States

IPD SHARING:
Plan to Share IPD: Undecided
Undecided where the research team would like to submit the article for publication